CLINICAL TRIAL: NCT05194917
Title: Aim-3: Alzheimer's Disease and Related Dementias Prevention Messaging to Increase Smoking Cessation Attempts in Older Adult Smokers
Brief Title: Motivating Change in Aging Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0650; K23AG067929 (NIH); A534252 (Other: UW Madison)
Record Dates: First submitted 2022-01-05; First posted 2022-01-18 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
Keywords: older smoker; motivational intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Older Smoker Motivational Intervention (Experimental): Message package focused on the link between smoking and dementia
  Interventions: Other: Older Smoker Motivational Intervention
- Control Motivational Message 1 (Active Comparator): CDC TIPS from former smokers campaign
  Interventions: Other: Control Motivational Message
- Control Treatment as Usual (No Intervention): No intervention
- Control Motivational Message 2 (Active Comparator): American Lung Association campaign
  Interventions: Other: Control Motivational Message

INTERVENTIONS:
Other: Older Smoker Motivational Intervention — OSMI identified in Aim 2 of the study, motivational interventions will be delivered via mailer with QR video code.
  Other Names: OSMI
  Arms: Older Smoker Motivational Intervention
Other: Control Motivational Message — One control motivational message with a standard health- and EBST access-related content (i.e., "Quitting smoking is the best thing you can do for your health. Call 1-800-QUIT-NOW for help."), motivational interventions will be delivered via mailer with QR video code.
  Arms: Control Motivational Message 1; Control Motivational Message 2

SUMMARY:
The purpose of this research is to evaluate messages that motivate older smokers to make quit attempts using evidence based smoking treatments (EBSTs). 200 participants will be recruited nationally (within the United States) primarily via social media advertisements. Participation will include up to 2 interviews by telephone and receiving flyers via mail.

DETAILED DESCRIPTION:
Overview. This study will use a pre-post design to assess feasibility and preliminary effectiveness of a developed Older Smoker Motivational Intervention (OSMI) presented in a large primary care clinic. Participants will be randomized to one of four messaging interventions; 1) active control (CDC TIPS from former smokers campaign), 2) active control (American Lung Association campaign), 3) treatment condition including message package focused on the link between smoking and dementia, 4) no intervention control. The messaging intervention will be delivered via mail, which will include a QR code link that will allow participants to view associated motivational video. Participants will then complete the first of 2 telephone survey assessments (lasting ~30 minutes). Participants will then receive three mailers over the next couple of months and will schedule their follow-up call approximately 2.5 months later. At one to two weeks, one month, and two months after this call they will be mailed the corresponding message to their group (no intervention group will not be sent a message package). Follow up telephone assessments will occur within approximately 1-2 weeks following intervention exposure marked by date the intervention mailer was sent.

Participants. Older adults from the community (N=200) who are ages 50-80, self-report being a current smoker, do not hold a current diagnosis of dementia or Mild Cognitive Impairment (MCI), can read and write in English will be eligible to participate, located within the United States.

Setting/Recruitment. Participants will be recruited nationally (within the United States) primarily via social media advertisements. Should these efforts fail, the investigators will use flyers and television advertisements. Those interested in participating in the study will call the provided contact information to enroll in the study directly with University of Wisconsin Center for Tobacco Research and Intervention (UW-CTRI) staff. Upon contacting UW-CTRI, the investigators will confirm their location via their provided address. All data collected for this study will be stored an a secure departmental server (electronic data) or in a locked file cabinet in a locked room at UW-CTRI (physical copies of data). Audio files of recordings will be stored on a secure departmental server.

Procedure and Assessments. Upon study initiation 200 participants will be recruited for the study and provide informed consent. After consent they will be randomized to one of the 4 study conditions (active control1, active control 2, no intervention, treatment condition). They will then complete the first of 2 telephone survey assessments (lasting ~25 minutes). Participants will then be informed they will receive three mailers over the next couple of months and will schedule their follow-up call approximately 2.5 months later. At two weeks, one month, and two months after this call they will be mailed the corresponding message to their group (no intervention group will not be sent a message package). Follow up telephone assessments will occur within approximately 1-2 weeks following intervention exposure marked by date the intervention mailer was sent. Up to 20 participants randomized to the intervention condition will complete an additional brief qualitative interview following their second telephone survey assessment (lasting ~20 minutes). The qualitative interview will focus on the perceived impact of the message, preferred number of message exposures, preferred modality of message receipt, and suggested improvement to message content. Health Believe Model (HBM)1 constructs assessed include: perceived severity, perceived benefits (i.e., efficacy of EBSTs; impact of quitting on Alzheimer's disease and related dementias (ADRD) risk), perceived barriers (i.e., knowledge of how to access EBSTs in healthcare setting), and self-efficacy (i.e., confidence in ability to quit in the next 30 days).

Analyses. The investigators will evaluate preliminary effectiveness by descriptively comparing primary (1) and secondary (2) outcomes longitudinally (baseline vs. follow up) within participants, as well as cross-sectionally comparing follow-up data by treatment randomization groups (Intervention Message vs. Control Message; Intervention Message vs. Treatment as Usual (TAU); TAU vs. Control Message). The investigators will assess feasibility during follow-up via receipt and comprehension of messages. The HBM1 outcomes will be compared longitudinally within participant to identify potential mechanisms of action for the interventions and identify potential changes to the interventions prior to a larger randomized controlled trial (RCT). Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) domains preliminarily assessed will include (1) Reach: comprehension of motivational and access message; (2) Efficacy on smoking-cessation related beliefs and intentions (i.e., motivation to quit, quit attempts, and use of EBSTs when quitting); and (3) Implementation of the novel OSMI will be assess via qualitative interviews with participants.

ELIGIBILITY:
Inclusion Criteria:

* ages 50-80
* can read and write English
* current smoker

Exclusion Criteria:

* current diagnosis of dementia or mild cognitive impairment

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne L Johnson, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Smoker Motivational Intervention (OSMI): Message package focused on the link between smoking and dementia
  Older Smoker Motivational Intervention: OSMI identified in Aim 2 of the study, motivational interventions will be delivered via mailer with QR video code.
- Control Motivational Message 1: CDC TIPS from former smokers campaign
  Control Motivational Message: One control motivational message with a standard health- and evidence based smoking treatments (EBST) access-related content (i.e., "Quitting smoking is the best thing you can do for your health. Call 1-800-QUIT-NOW for help."), motivational interventions will be delivered via mailer with QR video code.
Period: Overall Study
Arm/Group | Older Smoker Motivational Intervention (OSMI) | Control Motivational Message 1 | Control Treatment as Usual | Control Motivational Message 2
Started | 52 | 50 | 49 | 50
Completed | 45 | 45 | 43 | 45
Not Completed | 7 | 5 | 6 | 5
Not completed — Lost to Follow-up | 7 | 5 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Smoker Motivational Intervention | Control Motivational Message 1 | Control Treatment as Usual | Control Motivational Message 2 | Total
Number analyzed (Participants) | 52 | 50 | 49 | 50 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.92 (7.37) | 61.34 (6.33) | 62.53 (7.12) | 63.26 (7.41) | 62.52 (7.06)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 31 | 30 | 28 | 30 | 119
  Male | 21 | 20 | 20 | 20 | 81
  Non-binary | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 8 | 10 | 9 | 38
  White | 38 | 38 | 37 | 37 | 150
  More than one race | 2 | 1 | 2 | 2 | 7
  Unknown or Not Reported | 0 | 3 | 0 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 52 | 50 | 49 | 50 | 201

OUTCOME MEASURES:

1. Primary Outcome: Change in Motivation to Quit Within the Next 30 Days
Description: Motivation to Quit within the next 30 days is measured on a 10-point likert scale from 1 (not at all motivated) to 10 (extremely motivated); higher numbers indicate more motivation to quit.
Time Frame: baseline (during wave 1), up to 6 months (during wave 2)
Population: Several participants were lost to follow-up at 6 Months Post-Intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Smoker Motivational Intervention | Control Motivational Message 1 | Control Treatment as Usual | Control Motivational Message 2
Number analyzed (Participants) | 52 | 50 | 49 | 50
score on a scale
  Baseline Motivation to Quit within the next 30 days | 6.660 (2.225) | 6.10 (2.845) | 6.31 (2.852) | 6.34 (2.616)
  6 Months Post-intervention Motivation to Quit within the next 30 days: number analyzed (Participants) | 45 | 45 | 43 | 45
  6 Months Post-intervention Motivation to Quit within the next 30 days | 7.133 (2.4735) | 6.289 (2.9666) | 6.209 (2.9965) | 6.844 (2.8680)
  Change in Motivation to Quit within the next 30 days from Baseline to 6 Months Post-intervention: number analyzed (Participants) | 45 | 45 | 43 | 45
  Change in Motivation to Quit within the next 30 days from Baseline to 6 Months Post-intervention | -.6000 (2.30020) | -.4222 (2.91928) | -.1628 (3.28728) | -.3111 (2.06510)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected non-systematically by participant self-report at each telephone-based follow-up assessment through approximately 6 months months on study.
Description: Clinicaltrials.gov definitions were applied.
Arm/Group | Older Smoker Motivational Intervention | Control Motivational Message 1 | Control Treatment as Usual | Control Motivational Message 2
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT05194917/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT05194917/ICF_001.pdf